CLINICAL TRIAL: NCT06026137
Title: Use of the Efisiotrack System for Monitoring Prescribed Therapeutic Exercises in Patients With Shoulder Orthopedic Injuries in a Hospital Setting: a Pilot Feasibility Study
Brief Title: Use of the Efisiotrack System for Monitoring Patients With Shoulder Orthopedic Injuries
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Miguel Hernandez de Elche (Other)
Collaborators: Hospital General Universitario Elche (Other)
Responsible Party: Principal Investigator, JOSE VICENTE TOLEDO MARHUENDA, Principal Investigator, Universidad Miguel Hernandez de Elche
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JVT002
Record Dates: First submitted 2023-07-18; First posted 2023-09-06 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Shoulder Injuries
Keywords: rehabilitation; shoulder injury; monitoring device; adherence
MeSH Terms: conditions — Shoulder Injuries

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- eFisioTrack Group (Experimental): Use of the eFisioTrack platform in the experimental group to perform active exercises as part of their shoulder rehabilitation. These will. bee performed independently by each patient in a hospital room, using the efisioTrack system without supervision by the physiotherapist.
  The subjects will be previously instructed in the use of the system in two 20-minute sessions. The type of exercise and its parameters will be chosen and progressed considering the functional status of the patient and being similar to those executed under the physiotherapist's supervision.
  Interventions: Procedure: eFisioTrack Group
- Excercises Group (Active Comparator): Patients who performed the exercise program supervised by the physical physiotherapist in a hospital room.
  Interventions: Procedure: Excercises Group

INTERVENTIONS:
Procedure: eFisioTrack Group — Application of manual therapy and physical modalities together with completion of the exercise program for functional recovery of the upper extremity using the efisioTrack system without supervision by the physiotherapist.
  Arms: eFisioTrack Group
Procedure: Excercises Group — Application of manual therapy and physical modalities together with completion of the exercise program for functional recovery of the upper extremity supervised by the physical physiotherapist in a hospital room.
  Arms: Excercises Group

SUMMARY:
To evaluate the effect on clinical variables of monitoring exercises prescribed for shoulder injury rehabilitation with the eFisioTrack platform in patients of the Rehabilitation Service at University Hospital of Elche.

DETAILED DESCRIPTION:
Patients who be referred to the rehabilitation service of the University Hospital of Elche (Spain) for physiotherapy treatment (manual therapy, exercise, stretching, and electrotherapy) after suffering orthopedic injury or surgery in the shoulder joint complex will be considered for enrollment in the study.

Patients will performed the prescribed physical therapy treatment, at least three times per week in sessions of 45 minutes in the hospital setting (application of manual therapy and physical modalities as ultrasound, heat/cold, laser, magnetic field therapy) together with completion of the exercise program for functional recovery of the upper extremity (exercises for muscle strength, scapular stability, joint mobility, and proprioception).

Following baseline examination, patients will be randomly assigned to either physiotherapist-supervised exercise (control group) or monitoring by the eFisioTrack system (experimental group) to perform active exercises as part of their shoulder rehabilitation. These will be performed independently by each patient in a hospital room without supervision by the physiotherapist.

The following patient-reported outcome measures will be used to assess participants' shoulder pain and function: the Disabilities of Arm, Shoulder and Hand (DASH) score and the Constant-Murley (CM) score.

All participants will be assessed at baseline on their first visit to the physical therapy area and at one-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years old and be able to read and understand Spanish.
* Suffer a traumatic or degenerative shoulder injury, with or without surgical treatment.
* Have a prescription for rehabilitative physical therapy that includes active exercises.

Exclusion Criteria:

-Had a concomitant injury on an upper extremity or the cervical spine at the time of participation or sequelae of previous injuries in the area.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-06-29 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Disabilities of Arm, Shoulder and Hand (DASH) score | At baseline and at one month follow-up.
  DASH - Measures symptoms and degree of function related to a disorder in the upper extremity. The DASH Outcome Measure is scored in two components: the disability/symptom section (30 items, scored 1-5) and the optional high performance Sport/Music or Work section (4 items, scored 1-5). At least 27 of the 30 items must be completed for a score to be calculated. The assigned values for all completed responses are simply summed and averaged, producing a score out of five. This value is then transformed to a score out of 100 by subtracting one and multiplying by 25. This transformation is done to make the score easier to compare to other measures scaled on a 0-100 scale. A higher score indicates greater disability.

SECONDARY OUTCOMES:
Constant-Murley (CM) score. | At baseline and at one month follow-up.
  CMS - specific instrument for assessing the shoulder joint: pain; ability to perform daily activities; mobility and strength. The Constant-Murley score (CMS) is a 100-points scale composed of a number of individual parameters. These parameters define the level of pain and the ability to carry out the normal daily activities of the patient. The test is divided into four subscales: pain (15 points), activities of daily living (20 points), strength (25 points) and range of motion: forward elevation, external rotation, abduction and internal rotation of the shoulder (40 points). The higher the score, the higher the quality of the function.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Roses Conde, Ph, Study Director — Hospital Generalof Elche
Locations (1):
- Hospital General of Elche, Elche, Alicante, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Holmgren T, Bjornsson Hallgren H, Oberg B, Adolfsson L, Johansson K. Effect of specific exercise strategy on need for surgery in patients with subacromial impingement syndrome: randomised controlled study. BMJ. 2012 Feb 20;344:e787. doi: 10.1136/bmj.e787. PMID 22349588
- [Background] Baroni MP, Jacob MFA, Rios WR, Fandim JV, Fernandes LG, Chaves PI, Fioratti I, Saragiotto BT. The state of the art in telerehabilitation for musculoskeletal conditions. Arch Physiother. 2023 Jan 4;13(1):1. doi: 10.1186/s40945-022-00155-0. PMID 36597130
- [Background] Carbonaro N, Lucchesi I, Lorusssi F, Tognetti A. Tele-monitoring and tele-rehabilitation of the shoulder muscular-skeletal diseases through wearable systems. Annu Int Conf IEEE Eng Med Biol Soc. 2018 Jul;2018:4410-4413. doi: 10.1109/EMBC.2018.8513371. PMID 30441330
- [Background] Hervas MT, Navarro Collado MJ, Peiro S, Rodrigo Perez JL, Lopez Mateu P, Martinez Tello I. [Spanish version of the DASH questionnaire. Cross-cultural adaptation, reliability, validity and responsiveness]. Med Clin (Barc). 2006 Sep 30;127(12):441-7. doi: 10.1157/13093053. Spanish. PMID 17040628
- [Result] Lucas J, van Doorn P, Hegedus E, Lewis J, van der Windt D. A systematic review of the global prevalence and incidence of shoulder pain. BMC Musculoskelet Disord. 2022 Dec 8;23(1):1073. doi: 10.1186/s12891-022-05973-8. PMID 36476476
- [Result] Greenberg DL. Evaluation and treatment of shoulder pain. Med Clin North Am. 2014 May;98(3):487-504. doi: 10.1016/j.mcna.2014.01.016. Epub 2014 Mar 22. PMID 24758957
- [Result] Page MJ, Green S, McBain B, Surace SJ, Deitch J, Lyttle N, Mrocki MA, Buchbinder R. Manual therapy and exercise for rotator cuff disease. Cochrane Database Syst Rev. 2016 Jun 10;2016(6):CD012224. doi: 10.1002/14651858.CD012224. PMID 27283590
- [Result] Kromer TO, Tautenhahn UG, de Bie RA, Staal JB, Bastiaenen CH. Effects of physiotherapy in patients with shoulder impingement syndrome: a systematic review of the literature. J Rehabil Med. 2009 Nov;41(11):870-80. doi: 10.2340/16501977-0453. PMID 19841837
- [Result] Babatunde OO, Ensor J, Littlewood C, Chesterton L, Jordan JL, Corp N, Wynne-Jones G, Roddy E, Foster NE, van der Windt DA. Comparative effectiveness of treatment options for subacromial shoulder conditions: a systematic review and network meta-analysis. Ther Adv Musculoskelet Dis. 2021 Sep 9;13:1759720X211037530. doi: 10.1177/1759720X211037530. eCollection 2021. PMID 34527083
- [Result] Paraskevopoulos E, Plakoutsis G, Chronopoulos E, Maria P. Effectiveness of Combined Program of Manual Therapy and Exercise Vs Exercise Only in Patients With Rotator Cuff-related Shoulder Pain: A Systematic Review and Meta-analysis. Sports Health. 2023 Sep-Oct;15(5):727-735. doi: 10.1177/19417381221136104. Epub 2022 Dec 14. PMID 36517977
- [Result] Burns D, Boyer P, Razmjou H, Richards R, Whyne C. Adherence Patterns and Dose Response of Physiotherapy for Rotator Cuff Pathology: Longitudinal Cohort Study. JMIR Rehabil Assist Technol. 2021 Mar 11;8(1):e21374. doi: 10.2196/21374. PMID 33704076
- [Result] Eriksson L, Lindstrom B, Ekenberg L. Patients' experiences of telerehabilitation at home after shoulder joint replacement. J Telemed Telecare. 2011;17(1):25-30. doi: 10.1258/jtt.2010.100317. Epub 2010 Nov 12. PMID 21075802
- [Result] Carnevale A, Longo UG, Schena E, Massaroni C, Lo Presti D, Berton A, Candela V, Denaro V. Wearable systems for shoulder kinematics assessment: a systematic review. BMC Musculoskelet Disord. 2019 Nov 15;20(1):546. doi: 10.1186/s12891-019-2930-4. PMID 31731893
- [Result] Sliepen M, Lipperts M, Tjur M, Mechlenburg I. Use of accelerometer-based activity monitoring in orthopaedics: benefits, impact and practical considerations. EFORT Open Rev. 2020 Jan 28;4(12):678-685. doi: 10.1302/2058-5241.4.180041. eCollection 2019 Dec. PMID 32010456
- [Result] Rizzo JR, Thai P, Li EJ, Tung T, Hudson TE, Herrera J, Raghavan P. Structured Wii protocol for rehabilitation of shoulder impingement syndrome: A pilot study. Ann Phys Rehabil Med. 2017 Nov;60(6):363-370. doi: 10.1016/j.rehab.2016.10.004. Epub 2017 Mar 15. PMID 28330586
- [Result] Anwar N, Karimi H, Ahmad A, Gilani SA, Khalid K, Aslam AS, Hanif A. Virtual Reality Training Using Nintendo Wii Games for Patients With Stroke: Randomized Controlled Trial. JMIR Serious Games. 2022 Jun 13;10(2):e29830. doi: 10.2196/29830. PMID 35699989
- [Result] Adie K, Schofield C, Berrow M, Wingham J, Humfryes J, Pritchard C, James M, Allison R. Does the use of Nintendo Wii SportsTM improve arm function? Trial of WiiTM in Stroke: a randomized controlled trial and economics analysis. Clin Rehabil. 2017 Feb;31(2):173-185. doi: 10.1177/0269215516637893. Epub 2016 Jul 10. PMID 26975313
- [Result] Ruiz-Fernandez D, Marin-Alonso O, Soriano-Paya A, Garcia-Perez JD. eFisioTrack: a telerehabilitation environment based on motion recognition using accelerometry. ScientificWorldJournal. 2014 Jan 12;2014:495391. doi: 10.1155/2014/495391. eCollection 2014. PMID 24526898
- [Result] Tate AR, McClure PW, Young IA, Salvatori R, Michener LA. Comprehensive impairment-based exercise and manual therapy intervention for patients with subacromial impingement syndrome: a case series. J Orthop Sports Phys Ther. 2010 Aug;40(8):474-93. doi: 10.2519/jospt.2010.3223. PMID 20710088
- [Result] Franchignoni F, Vercelli S, Giordano A, Sartorio F, Bravini E, Ferriero G. Minimal clinically important difference of the disabilities of the arm, shoulder and hand outcome measure (DASH) and its shortened version (QuickDASH). J Orthop Sports Phys Ther. 2014 Jan;44(1):30-9. doi: 10.2519/jospt.2014.4893. Epub 2013 Oct 30. PMID 24175606
- [Result] Roy JS, MacDermid JC, Woodhouse LJ. A systematic review of the psychometric properties of the Constant-Murley score. J Shoulder Elbow Surg. 2010 Jan;19(1):157-64. doi: 10.1016/j.jse.2009.04.008. PMID 19559630
- [Result] Kitis A, Celik E, Aslan UB, Zencir M. DASH questionnaire for the analysis of musculoskeletal symptoms in industry workers: a validity and reliability study. Appl Ergon. 2009 Mar;40(2):251-5. doi: 10.1016/j.apergo.2008.04.005. Epub 2008 Jun 16. PMID 18555973
- [Result] Pastora-Bernal JM, Martin-Valero R, Baron-Lopez FJ, Moyano NG, Estebanez-Perez MJ. Telerehabilitation after arthroscopic subacromial decompression is effective and not inferior to standard practice: Preliminary results. J Telemed Telecare. 2018 Jul;24(6):428-433. doi: 10.1177/1357633X17706583. Epub 2017 Apr 27. PMID 28449618
- [Result] Correia FD, Molinos M, Luis S, Carvalho D, Carvalho C, Costa P, Seabra R, Francisco G, Bento V, Lains J. Digitally Assisted Versus Conventional Home-Based Rehabilitation After Arthroscopic Rotator Cuff Repair: A Randomized Controlled Trial. Am J Phys Med Rehabil. 2022 Mar 1;101(3):237-249. doi: 10.1097/PHM.0000000000001780. PMID 33935152
- [Result] Grassi FA, Tajana MS. The normalization of data in the Constant-Murley score for the shoulder. A study conducted on 563 healthy subjects. Chir Organi Mov. 2003 Jan-Mar;88(1):65-73. English, Italian. PMID 14584318
- [Result] Kachingwe AF, Phillips B, Sletten E, Plunkett SW. Comparison of manual therapy techniques with therapeutic exercise in the treatment of shoulder impingement: a randomized controlled pilot clinical trial. J Man Manip Ther. 2008;16(4):238-47. doi: 10.1179/106698108790818314. PMID 19771196

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-07-17): https://cdn.clinicaltrials.gov/large-docs/37/NCT06026137/Prot_SAP_ICF_000.pdf